CLINICAL TRIAL: NCT02254564
Title: PCR (Polymerase Chain Reaction) Assay for Diagnosis of Sarcoptes Scabiei
Status: Completed | Type: Observational
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Principal Investigator, Dayna Diven, Physician, Seton Healthcare Family
Other Study IDs: Scabies 1
Record Dates: First submitted 2014-09-29; First posted 2014-10-02 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-06

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Superficial skin scrapings scales that are collected on microscope slides, which are used to determine diagnosis in clinical settings. After clinicians view the slide under the microscope, the slide is then discarded.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Positive Scrapings: Skin scrapings that are positive for scabies
- Negative Controls: collect negative controls from patients in whom tinea (superficial fungal infection) was clinically suspected. Samples from patients with demodex folliculitis (a mite that is commonly found in oil glands on the face) are also intended to be used as negative controls as well.

SUMMARY:
The main objective of this study is to identify unique DNA sequences within the genome of human scabies that can be utilized to identify the parasite through PCR.

DETAILED DESCRIPTION:
The main objective of this proposed study is to identify unique DNA sequences within the genome of human scabies that can be utilized to identify the parasite through polymerase chain reaction or PCR. The goal of the project is to design an assay that can distinguish samples from skin scrapings containing scabies mites, eggs, or fecal material confirmed by clinic based microscopic evaluation (gold standard) from negative controls (i.e. scrapings for tinea and/or demodex folliculitis) that do not contain Sarcoptes scabiei. We hypothesize that specifically amplifying the unique regions of the Scabies genome using PCR can serve as a means to diagnosis infestations in humans. To address this question, we will optimize PCR amplification of known scabies samples then apply our procedure to DNA extracted from patient samples.

ELIGIBILITY:
Inclusion Criteria:

* 1. Male/Female of all ages whose standard clinical treatment produces one or more of the following:

  * Slides from skin scrapings containing scabies mites, eggs, and/or fecal material
  * Slides from skin scrapings of suspected tinea
  * Slides from skin scrapings of demodex mites

Exclusion Criteria:

* 1. Patients who are clinically concerning for having both scabies and tinea/demodex folliculitis to avoid contamination of positive and negative controls in the same sample. Subjects or guardians who cannot understand and read English and so are unable to consent to participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be recruited upon identifying of scabies by microscopy or when a scraping is performed for suspected tinea or demodex folliculitis
Sampling Method: Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Identification of DNA sequences within scabies that can be used to identify the parasite through PCR | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Dayna Diven, MD, Principal Investigator — Seton Healthcare Family
Locations (5):
- United States (5):
  - Seton Family of Hospitals- Trinity and Hays Clinic, Austin, Texas
  - University Medical Center Brackenridge and Paul Bass Clinic, Austin, Texas
  - University of Texas Physicians at Trinity, Austin, Texas
  - Seton Family of Hospitals- Dell Children's Medical Center of Central Texas and Specially for Children, Austin, Texas
  - Seton Family of Hospitals- Seton Luling Family Medicine Clinic and Lockhart Specialty Clinic, Lockhart, Texas

IPD SHARING:
Plan to Share IPD: No